CLINICAL TRIAL: NCT02483091
Title: Chiropractors Can Do: Testing the Feasibility of Intervening to Optimize Chiropractic Care for Adults With Neck Pain Disorders: A Pilot Cluster Randomized Controlled Trial
Brief Title: Testing the Feasibility of Intervening to Optimize Chiropractic Care for Adults With Neck Pain Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Andre Bussieres, Assistant Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: G241013 R.E Strauss X-C 218563
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Neck Pain
Keywords: Knowledge translation; Clinical practice guidelines; Multimodal care; Brief Action Planning; Feasibility outcomes
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multifaceted KT intervention (Experimental): Webinars, online vignettes and e-module, copy of guideline recommendations
  Interventions: Behavioral: Multifaceted KT intervention
- Control (No Intervention): Printed copy of guideline recommendations

INTERVENTIONS:
Behavioral: Multifaceted KT intervention — The intervention consists of three webinars followed by the quiz, two online case scenario and a video on BAP model plus a printed copy of Clinical Practice Guideline (CPGs) on NSNP.
  After completing these modules and learning the key strategies, each chiropractor will recruit five neck pain patients and implement the strategies on their patients to measure the clinical outcomes for a follow-up of three months.
  The control group will receive only a printed copy of CPGs. A checklist of proxy measures embedded within patient encounter forms will be used to assess chiropractors' compliance with guideline recommendations at study onset and at three months.
  Arms: Multifaceted KT intervention

SUMMARY:
To assess the feasibility of conducting a larger cluster randomized controlled trial to facilitate the effectiveness of a complex Knowledge Translation (KT) intervention, i.e. implementation of multimodal care, into chiropractic clinical practice, designed to improve the management of patients with Non-Specific Neck Pain (NSNP) disorders.

To evaluate feasibility, the investigators will ascertain how well participating chiropractors and patients adhere to the study protocol and will solicit feedback from them about the overall usefulness of the content and format of the KT intervention. This study will determine planning for the main study and also the outcomes to be used as a primary outcome.

DETAILED DESCRIPTION:
The aim of this pilot study project is to determine the feasibility of implementing a multifaceted KT intervention to promote the use of multimodal care by chiropractors managing patients with NSNP.

Design: Cluster randomized controlled pilot and feasibility trial. Chiropractors in private practice in Canada will be randomized to receive either a theory-based tailored KT intervention in the experimental group or simply a printed copy of the guideline in the control group.

Study population and sample size: 30 chiropractors will be recruited from a random, nationally representative sample of 200 chiropractors. Each chiropractor will recruit five neck pain patients for a total of 150 patients.

The design of the KT intervention was informed by the results of a related qualitative study (Theoretical Domains Framework interviews) and consists of a series of three webinars, two online case scenarios, a self-management video on Brief Action Planning (BAP) and a printed copy of the practice guideline (Bussières et al., 2015).

Primary feasibility outcomes for both chiropractors and patients include rates of: 1) recruitment, 2) study retention, and 3) adherence to the intervention (Tickle-Degnen, 2013). A checklist of proxy measures embedded within patient encounter forms will be used to assess chiropractors' compliance with guideline recommendations e.g., exercise and self-care prescriptions, at study onset and at three months follow-up.

Secondary outcomes include whether or not the chiropractor's recommended multimodal care, scores on measures of behavioural constructs e.g., self-efficacy, knowledge.

Primary clinical outcomes for patients includes measures of pain intensity and neck pain-specific disability.

Analyses from this pilot study will focus on generating point estimates and corresponding 95% confidence intervals for parameters of a priori interest (e.g., recruitment, retention, adherence, pain intensity, neck disability index).

Discussion: The main strength of this study includes its use of a representative sample and randomized controlled design. The results of this study will inform the design of a larger cluster randomized controlled trial aimed at confirming the effectiveness and increasing the use of multimodal care by chiropractors managing patients with NSNP.

ELIGIBILITY:
Chiropractors

Inclusion criteria:

* Registered with their professional licensing boards and in private practice in the Canada;
* Graduated at least one year ago;
* Provide chiropractic treatment to a minimum of two adults (age 18-65) with neck pain per week;
* Speak English or French; and
* Have access to Internet.

Exclusion criteria:

* Chiropractors will be excluded if they have already attended the webinar series or the self-management learning module. Prior webinar and learning module participants will have needed to register beforehand, which therefore provides the mechanism for confirming study ineligibility.

Patients

Inclusion criteria:

* Attend a consenting chiropractor for non-specific neck pain of any duration;
* Aged between 18 and 65, with a primary complaint of acute (<3 months) or chronic (>3 months) neck pain presenting as a new condition for treatment at the participating clinic;
* Fluency in English or French to a level where they can read and understand the study information sheet, complete the consent form, and respond to the telephone-administered questionnaire. This will be assessed by the staff member of each chiropractor's team at the time of screening; and
* Provide written informed consent.

Exclusion criteria:

* Previous neck surgery;
* Presence of Red flags;
* Pregnancy; and
* Chiropractic care received in the preceding 3 months for a complaint of neck pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome (composite outcome measure) | 6 months
  The main outcome of interest is feasibility that includes recruitment, retention, adherence to the study protocol and effectiveness potential.
  Recruitment rate include: 1) eligibility rate (number of eligible chiropractors and patients divided by invited chiropractors or patients) and 2) participation rate (number agreeing to participate divided by eligible chiropractors or patients).
  Retention rate: Number of chiropractors and patients who completed all outcome measures at baseline and at 3 month follow-up plus rate of completion of questionnaires by chiropractors (measures of behavioural constructs) and patients (clinical outcomes).
  For chiropractors, rate of adherence includes attendance of all 3 webinars, associated quizzes, 2 clinical vignettes and the self-management learning module; For patients, rate of adherence includes follow-up visits, prescribed home exercise and physical activity.

SECONDARY OUTCOMES:
Scores on measures of behavioural constructs (composite outcome measure) | 6 months
  For chiropractors: Scores on measures of behavioural constructs (levels of knowledge and self-efficacy) for recommended multimodal care.

OTHER OUTCOMES:
Pain | 3 months (before and at the end of treatment)
  Self-rated level of pain on an 11 points continuous Visual Analogue Scale (VAS)
Disability | 3 months (before and at the end of treatment)
  Self-rated disability due to neck pain measured on the Neck Disability Index (NDI). Scale range and subscales:10 items in total, each item is scored from 0-5 ("0" = no disability and "5" = full disability) for a total of 50
Satisfaction with care | 3 months (end of treatment) and 3 months of follow-up
  Self-rated satisfaction with care measured on the Short Form Patient Satisfaction Questionnaire (PSQ-18). Scale range and subscales:10 items in total, each item is scored from 1-5 ("1" = strongly agree and "5" = strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: André E Bussières, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bussieres AE, Al Zoubi F, Quon JA, Ahmed S, Thomas A, Stuber K, Sajko S, French S; Members of Canadian Chiropractic Guideline Initiative. Fast tracking the design of theory-based KT interventions through a consensus process. Implement Sci. 2015 Feb 11;10:18. doi: 10.1186/s13012-015-0213-5. PMID 25880218
- [Background] Tickle-Degnen L. Nuts and bolts of conducting feasibility studies. Am J Occup Ther. 2013 Mar-Apr;67(2):171-6. doi: 10.5014/ajot.2013.006270. PMID 23433271
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Derived] Dhopte P, French SD, Quon JA, Owens H, Bussieres A; Canadian Chiropractic Guideline Initiative. Guideline implementation in the Canadian chiropractic setting: a pilot cluster randomized controlled trial and parallel study. Chiropr Man Therap. 2019 Jul 17;27:31. doi: 10.1186/s12998-019-0253-z. eCollection 2019. PMID 31346409
- [Derived] Dhopte P, Ahmed S, Mayo N, French S, Quon JA, Bussieres A. Testing the feasibility of a knowledge translation intervention designed to improve chiropractic care for adults with neck pain disorders: study protocol for a pilot cluster-randomized controlled trial. Pilot Feasibility Stud. 2016 Jul 20;2:33. doi: 10.1186/s40814-016-0076-9. eCollection 2016. PMID 27965852